CLINICAL TRIAL: NCT01607723
Title: Comparison of Two New Ventilatory Modes: NAVA vs PAV+: a Randomized Controlled Cross-over Study: the "NAVA-PAV" Study
Brief Title: "NAVA-PAV" Study: a Cross-over Comparative Study of 2 Advanced Modes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: UF 8916
Record Dates: First submitted 2012-04-18; First posted 2012-05-30 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Critical Illness; Mechanical Ventilation; Intensive Care; Ventilation Weaning
Keywords: Sleep pattern; Mechanical ventilation; weaning; Intensive Care; NAVA (Neurally Adjusted Ventilatory Assist); PAV+ (Proportional Assist Ventilation Plus)
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- NAVA ventilatory mode (Other)
  Interventions: Other: NAVA ventilatory mode
- PAV+ ventilatory mode (Other)
  Interventions: Other: PAV+ ventilatory mode

INTERVENTIONS:
Other: NAVA ventilatory mode — The two ventilatory modes will be studied during 24h in intubated patients in random order.
  Arms: NAVA ventilatory mode
Other: PAV+ ventilatory mode — The two ventilatory modes will be studied during 24h in intubated patients in random order.
  Arms: PAV+ ventilatory mode

SUMMARY:
Neurally adjusted ventilatory assist (NAVA) and Proportional Assist Ventilatory Plus (PAV +) are new modes of mechanical ventilation that delivers ventilatory assist in proportion to the electrical activity of the diaphragm for NAVA and to patients efforts for PAV +. The goal of this trial is to compare oxygenation,ventilator comfort, patients -ventilator asynchronies, and sleep pattern between NAVA and PAV+.

DETAILED DESCRIPTION:
Twenty patients will be enrolled. They will be ventilated with PAV+ and NAVA for one day, each in a randomized crossover order. The oxygenation,ventilator comfort, patients -ventilator asynchronies, and sleep pattern will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Estimated remaining duration of mechanical ventilation for more than two days
* patient alert and calm
* Surrogate decision maker's consent

Exclusion Criteria:

* Clinical contraindication for the use of NAVA: contraindications for an EAdi catheter placement (e.g., esophageal varices, upper gastrointestinal bleeding, gastroesophageal surgery)
* Clinical instability for any reason
* Contraindications for continuing intensive care treatment
* Patient under tutelage
* Age < 18 years
* Pregnancy
* No French health insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-05; Primary Completion 2012-05 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Oxygenation in NAVA and in PAV+ | after one day of ventilation in NAVA and in PAV+

SECONDARY OUTCOMES:
Ventilatory comfort | Every 6 hours in the two ventilatory modes
  Ventilatory comfort will be assessed by :
  * objective criteria expressed in time spent in each mode in the area called "comfort" (12 < Respiratory frequence < 28 c/min ; Current Volume > 300 mL and EtCO2 < 55 mmHg)
  * subjective criteria expressed by the self-assessment of the patient's comfort on a visual analogic scale.
Patient-ventilator asynchronies | During the 24h of mechanical ventilation in NAVA and in PAV+
  The patient-ventilator asynchronies will be assessed by the asynchronie index (number of asynchronies / number of respiratory cycles). The number of asynchronies will be assessed by the investigator, on the records of the pression curves and the respirator outputs.
Ventilatory parameters | During the 24h of mechanical ventilation in NAVA and in PAV+
  The aeration and pulmonary ventilation will be assessed by electrical impedance (PulmoVista®500, Drager, Suisse).
Sleep pattern | During 24h of mechanical ventilation in NAVA and in PAV+

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology & Critical Care, St Eloi University Hospital, Montpellier, France